CLINICAL TRIAL: NCT06115551
Title: Cellular Effects of Fasting Mimicking Diet In Humans: An Interventional, Randomized, Open Label, Parallel Assignment Study
Brief Title: Fasting Mimicking Diet and Autophagy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L-Nutra Inc (Industry)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LNT22-017
Record Dates: First submitted 2023-10-20; First posted 2023-11-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Diet; Autophagy
Keywords: Fasting mimicking diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Subjects in the control group will be asked to keep their normal diet during the study period.
- FMD1-ProLon (Experimental): Subjects in FMD1 groups will be provided and asked to consume a 5-day low calorie fasting-mimicking diet (ProLonTM).
  Interventions: Combination Product: Fasting Mimicking Diet
- FMD2-ProMete (Experimental): Subjects in FMD2 groups will be provided and asked to consume a 5-day low calorie fasting-mimicking diet (ProMeteTM).
  Interventions: Combination Product: Fasting Mimicking Diet

INTERVENTIONS:
Combination Product: Fasting Mimicking Diet — FMD is a 5-day low calorie fasting-mimicking diet.
  Other Names: ProLon, ProMete
  Arms: FMD1-ProLon; FMD2-ProMete

SUMMARY:
This study aims to evaluates autophagy in circulating white blood cells from generally healthy human volunteers exposed to fasting mimicking diet (FMD), a 5-day dietary regimen.

DETAILED DESCRIPTION:
Fasting-mimicking diet (FMD) was developed to mimic the endocrine and metabolic effects that water-only fasting, while providing a modest calories and essential nutrients. The health benefits of FMD are caused by several molecular mechanisms, including the reduction of body weight, ectopic fat storage, insulin levels, endogenous glucose production and IGF-1. Autophagy is a catabolic membrane-trafficking phenomenon observed in yeast and mammalian cells. Nutrient deprivation induces autophagy. Autophagy has been proposed to be a fundamental cellular process being linked to aging and the progression of age-related diseases. The objective of this study is to evaluate the effects of consuming two FMD formulations on the autophagy process in the cell.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent;
* Ability and willingness to perform the study tests and adhere to study protocol (to the best of the participant's knowledge);
* BMI 20-35 kg/m2 (inclusive) at screening;

Exclusion Criteria:

* Diabetes treatment other than diet or metformin monotherapy;
* History of gastric bypass;
* Subjects with recent weight loss (>5%), use of weight loss medication, participated in a weight loss program in the past 3 months;
* Type 1 diabetes (based on medical history provided at screening);
* Use of immune suppression drugs;
* Contraindication for study foods (special food needs and allergy);
* Women who are pregnant;
* Alcohol dependency (alcohol intake greater than two drinks per day for women and three drinks per day for men).
* Has any medical disease or condition that, in the opinion of the principal investigator (PI) or appropriate study personnel, precludes study participation* (*Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial);

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Autophagy flux | Baseline to day 8
  PBMCs will be prepared with or without Chloroquine (autophagy flux inhibitor). LC3BI to LC3BII conversion, the lipidation of MAP1LC3B/LC3B (microtubule-associated protein 1 light chain 3 β), in the PBMCs will be accessed by western blot.
  Autophagy-dependent degradation of SQSTM1/p62, a receptor and scaffold protein interacting with LC3 and ubiquitinated proteins, will be accessed by western blot.

SECONDARY OUTCOMES:
Metabolomic change | Baseline to day 8
  Plasma will be analyzed by high throughput RNA sequencing for gene expression changes.
Autophagy-related gene expression | Baseline to day 8
  PBMCs will be prepared with or without Chloroquine (autophagy flux inhibitor). PBMC RNA samples will be analyzed using ultra high-performance liquid chromatography/tandem accurate mass spectrometry (UHPLC/MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Espinoza, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Espinoza SE, Park S, Connolly G, Qi W, Zhang N, Semwal M, Li Y, Lauzon M, Salmon AB, Hsu W, Wei M, Musi N. Effect of fasting-mimicking diet on markers of autophagy and metabolic health in human subjects. Geroscience. 2025 Dec 11. doi: 10.1007/s11357-025-02035-4. Online ahead of print. PMID 41372565